CLINICAL TRIAL: NCT02603653
Title: Cognitive Sequels of Cushing Syndrome
Brief Title: Assessment of Persistent Cognitive Impairment After Cure of Cushing's Disease
Acronym: MEMOCUSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Purpose: Diagnostic
Other Study IDs: C15-02; IDRCB (Registry Identifier: 2015-A00617-42)
Record Dates: First submitted 2015-11-03; First posted 2015-11-13 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2015-11

CONDITIONS: Cushing's Disease
MeSH Terms: conditions — Pituitary ACTH Hypersecretion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients (Experimental): Virtual radial task in 3D
  Interventions: Device: Virtual radial task in 3D
- Controls (Experimental): Virtual radial task in 3D
  Interventions: Device: Virtual radial task in 3D

INTERVENTIONS:
Device: Virtual radial task in 3D — The virtual radial task is a labyrinth in 3D with twelve ways. The primary aim of our study is the evaluation of persistent cognitive impairments (hippocampal memory) according to the responses of participants after instructions to choose the right way in the labyrinth.

SUMMARY:
Cushing's disease is a state of chronic endogenous glucocorticoid excess. Cushing's disease is responsible for increased morbidity and mortality. Recent studies have pinpointed the frequency of somatic sequelas and persistent alteration in quality of life despite the cure of the disease. More specifically, a few studies have described persistent psychopathology, maladaptive personality and cognitive impairments in patients with a history of Cushing's disease. Among these, hippocampal memory deficits have been found in the majority of studies, a finding that is consistent with the alterations described in hippocampal neurons during chronic exposure to glucocorticoids. However, the tools currently available to assess hippocampal-dependent memory are multiple, sometimes difficult to perform by clinicians and to analyze or may lack of diagnostic sensitivity. The investigators have recently developed an original tool, the virtual radial task in 3D, which has shown to be reliable to detect subtle alterations in hippocampal-dependent memory in several human diseases. The primary aim of the study is the evaluation of persistent cognitive impairments (hippocampal memory) in patients cured of Cushing's disease for at least one year using the virtual radial task in 3D and to compare it with that obtained with classical cognitive tests.

ELIGIBILITY:
Inclusion Criteria:

Patients :

* history of Cushing's Disease
* aged : 18 - 60 years
* Biological remission of Cushing's disease for at least one year
* Affiliation to Social Security
* Informed consent signed by patient and investigator (at the latest the inclusion's day, before study's exams)

For controls :

* People aged 18 to 60 years matched to patients for age, sex and educational level
* Affiliation to Social Security
* Informed consent signed by patient and investigator (at the latest the inclusion's day, before study's exams)

Exclusion Criteria:

For patients :

* Persistent hypercortisolism (even mild)
* Current treatment of hypercortisolism with drugs
* Obesity (BMI >30 kg/m²)
* Alcohol or drug addiction present or past
* Growth hormone deficit
* Diabetes mellitus with hemoglobin A1c > 7.5% and/or fasting blood glucose > 1.4 g/L
* History of pituitary radiotherapy
* History of cerebrovascular or neuro-cerebral disease
* untreated dysthyroidism
* Current psychotropic drug treatment
* Pregnancy
* Use of glucocorticoids in the last 3 months before study (aside hydrocortisone replacement therapy)
* Excessive hydrocortisone replacement therapy (unadjusted to weight and/or with evening administration)

For controls :

* Obesity (BMI >30 kg/m²)
* Alcohol or drug addiction present or past
* Current psychotropic drug treatment
* History of cerebrovascular or neuro-cerebral disease
* Current pregnancy
* Chronical use of corticoid (> 1 month), current or past
* Use of glucocorticoids in the last 3 months before study (aside hydrocortisone replacement therapy)
* Diabetes mellitus with hemoglobin A1c > 7.5% and/or fasting blood glucose > 1.4 g/L
* Obesity (BMI >30 kg/m²)
* untreated dysthyroidism

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02-04 (Actual); Primary Completion 2017-02-12 (Actual); Study Completion 2017-08-03 (Actual)

PRIMARY OUTCOMES:
Percentage of right answers at virtual radial task in 3D | baseline
  Comparison of right answers in patients cured of Cushing's disease and in controls.

SECONDARY OUTCOMES:
General Quality of life | baseline
  Comparison of quality of life of patients and controls with validated general questionnaire : SF-36 (SF for Short Form health survey)
Specific Quality of life for Cushing's Disease | baseline
  Comparison of quality of life of patients and controls with validated specific questionnaire for Cushing's Disease : Cushing-QoL
Number of participants with anxiety | baseline
  Evaluation of anxiety in the two groups with Hospital Anxiety and Depression Scale (HADS) scale (questionnaire)
Number of participants with depression with MADRS | baseline
  Evaluation of depression in the two groups with Montgomery and Asberg Depression Rating Scale (MADRS) (questionnaire)
Number of participants with depression with HADS | baseline
  Evaluation of depression in the two groups with Hospital Anxiety and Depression Scale (HADS) scale (questionnaire)
Intensity of Cushing's syndrome | baseline
  Intensity of Cushing's disease will be evaluated with mean of free urinary cortisol. Hypothesis : intensity of hypercortisolism is correlated with sequels after cure.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Tabarin, Pr, Principal Investigator — Hôpital Haut Lévêque - Pessac (France)
Locations (1):
- Hôpital du Haut-Lévêque, Pessac, France

REFERENCES:
- [Result] Pupier E, Santos A, Etchamendy N, Lavielle A, Ferriere A, Marighetto A, Resmini E, Cota D, Webb SM, Tabarin A. Impaired quality of life, but not cognition, is linked to a history of chronic hypercortisolism in patients with Cushing's disease in remission. Front Endocrinol (Lausanne). 2022 Aug 8;13:934347. doi: 10.3389/fendo.2022.934347. eCollection 2022. PMID 36004342